CLINICAL TRIAL: NCT05136456
Title: A Phase II Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of SHR1459 Tablets in the Treatment of Primary Membranous Nephropathy (PMN)
Brief Title: Evaluate the Efficacy and Safety of SHR1459 Tablets in Patients With Primary Membranous Nephropathy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Reistone Biopharma Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RSB20926
Record Dates: First submitted 2021-11-17; First posted 2021-11-29 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Primary Membranous Nephropathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SHR1459 Low Dose (Active Comparator): Drug: SHR1459 SHR1459 oral 24weeks
  Interventions: Drug: SHR1459 Low Dose
- SHR1459 High Dose (Active Comparator): Drug: SHR0302 SHR1459 oral 24 weeks
  Interventions: Drug: SHR1459 High Dose
- Placebo (Placebo Comparator): Drug: Placebo Placebo oral 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SHR1459 Low Dose — SHR1459 oral tablets taken once daily (QD) for 24weeks
  Arms: SHR1459 Low Dose
Drug: SHR1459 High Dose — SHR1459 oral tablets taken once daily (QD) for 24 weeks
  Arms: SHR1459 High Dose
Drug: Placebo — Placebo oral tablets taken once daily (QD) for 24 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of SHR1459 tablets in patients with primary membranous nephropathy.

DETAILED DESCRIPTION:
This study is a phase II study to evaluate the efficacy and safety of SHR1459 tablets in patients with primary membranous nephropathy.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of primary membranous nephropathy based on renal biopsy before or during screening
2. Have not received any previous immunosuppressive therapy for primary membranous nephropathy or relapse after the treatment has achieved complete or partial remission (comprehensive judgment and recording by the investigator)
3. PLA2R-Ab titer ≥20RU/mL at screening
4. 24-hour urinary protein ≥ 3.5g/d at screening
5. Have eGFR ≥ 60 mL/min/1.73 m2 (based on CKD-EPI formula) at screening

Exclusion Criteria:

1. Any clue for coexist of secondary membranous nephropathy from medical records, laboratory tests or kidney biopsy
2. Existence of clinically significant infection within 1 month before screening,
3. Severe or not well controlled other complications
4. Abnormal in white blood cell count, neutrophil count, lymphocyte count or platelet count at screening, which were considered unfit for participating judged by investigators
5. ALT > 2 times ULN and/or AST > 2 times ULN and/or bilirubin >2 times ULN at screening
6. Subject has evidence of active, latent, or inadequately treated infection with Mycobacterium tuberculosis
7. Positive of hepatitis B surface antigen, hepatitis C antibody, HIV antibody or syphilis antibody at screening;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2023-08-28 (Estimated); Study Completion 2024-03-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects achieving complete or partial remission at week 24 | 24 Weeks
  Proportion of subjects achieving complete or partial remission at week 24

CONTACTS AND LOCATIONS:
Locations (19):
- China (19):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Zhongshan Hospital Xiamen University, Xiamen, Fujian
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Jiangsu Province People's Hospital, Nanjing, Jiangsu
  - Zhongda Hospital affiliated to Southeast University, Nanjing, Jiangsu
  - Subei People's Hospital of Jiangsu province, Yangzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Second Hospital of Jilin University, Changchun, Jilin
  - The First Affiliated Hospital of Baotou Medical College, Baotou, Nei Monggol
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Renji Hospital Shanghai Jiaotong University School of Medicine, Shanghai
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Tongji Hospital of Tongji University, Shanghai
  - Xinhua Hospital Affiliated To Shanghai Jiao Tong University School Of Medicine, Shanghai